CLINICAL TRIAL: NCT01272609
Title: Treatment of Port Wine Stains in Children With Pulsed Dye Laser and Timolol Gel
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-PP-11; 2010-022440-20 (EudraCT Number)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2011-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP + Timolol (Experimental): Three sessions of LCP in 595 nm (diameter of spot 7mm; duration of shooting 1,5 ms; Fluence 8 J / cm ²if LCP of Candela © or 7 J / cm ² if LCP of Cynosure ©) spaced out of 1 month. Twice-daily applications on the zone treated by the LCP of timolol frost and will be begun that very evening by the first session and will be pursued 15j after the 3rd session of LCP. The maximum surface of treatment will be 100 cms ².
  Interventions: Drug: Timolol + LCP
- LCP (Active Comparator): Three sessions of LCP in 595 nm (diameter of spot 7mm; duration of shooting 1,5ms; Fluence 8 J / cm ² if LCP of Candela © or 7 J / cm ² if LCP of Cynosure © spaced out of 1 month.
  Interventions: Device: LCP

INTERVENTIONS:
Drug: Timolol + LCP — Three sessions of LCP in 595nm (diameter of spot 7mm; duration of shooting 1,5ms; Fluence 8 J / cm ² if LCP of Candela © or 7 J / cm ² if LCP of Cynosure ©) spaced out of 1 month. Twice-daily applications on the zone treated by the LCP of timolol frost and will be begun that very evening by the first session and will be pursued 15j after the 3rd session of LCP. The maximum surface of treatment will be 100 cms ².
  Arms: LCP + Timolol
Device: LCP — Three sessions of LCP in 595nm (diameter of spot 7mm; duration of shooting 1,5ms; Fluence 8 J / cm ²if LCP of Candela © or 7 J / cm ²if LCP of Cynosure © spaced out of 1 month.
  Arms: LCP

SUMMARY:
Pulsed dye laser (PDL)is the gold standard treatment of port wine stains (PWS). However, many sessions are required and failure or relapses are not uncommon. It has been demonstrated that a neoangiogenesis occurs after PDL, explaining at least partially those failure. The objective of this study is to evaluate the use of a topical beta-blocker (timolol 1% gel) as a combination treatment with PDL for treating PWS.

Methods. Prospective multicenter study comparing PDL alone to PDL + timolol. Sessions of PDL will be performed once a month for 3 months. One group will be treated with PDL alone and the other will also applied timolol 1% gel twice a day during treatment. The evaluation will be done one month after the third session.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 months to 18 year-old.
* PWS of the face
* No prior treatement with PDL
* Membership or beneficiary of a national insurance scheme.
* Consent signed by the parents and by the patient if he is old enough to understand

Exclusion Criteria:

* Child with whom the angioma plan was already handled by laser or pulsed lamp
* Histories of asthma or obstructive bronchitis
* severe allergic Rhinitis and hyper bronchial ability to react
* Bradycardie sinusale, block auriculo-ventriculaires of the second or third degree
* unchecked Cardiac insufficiency
* cardiogenic Shock
* untreated Phéochromocytome
* Sentimentality in the timolol or in one of these excipients, and\or in the other bétabloquants
* Taken by floctafénine or by sultopride
* Taken of bétabloquants by oral route, of inhibitors calcic or of amiodarone
* severe peripheral circulatory Disorders(Confusions of Raynaud)
* arterial Low blood pressure
* Pregnancy and feeding
* Absence of effective contraception at the girls old enough to procreate
* Contraindication in the use of cream with lidocaïne and with prilocaïne

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
IGA | one month after the third session
  * IGA (investigator global assessment) at 3 or 4 marked improvement or complete clearance one month after the third session. Blinded evaluation by two physicians on standardized photos
  * Colorimetric analysis

SECONDARY OUTCOMES:
Subjective evaluation of the patients on visual analogical scale | three months
  Subjective evaluation of the patients on visual analogical scale

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Thierry, Pu-Ph, Principal Investigator — CHU de Nice - Service de Dermatologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (10):
- France (10):
  - CHU de Nice - 4 avenue Reine Victoria, Nice, Alpes-Maritimes
  - CHU de Bordeaux, Bordeaux
  - Hôpital Sévigné, Cesson-Sévigné
  - CHU de Dijon, Dijon
  - Clinique de Turin, Paris
  - CH de Quimper, Quimper
  - CHU de reims, Reims
  - Clinique Mathilde, Rouen
  - CHU de Touloluse, Toulouse
  - Clinique Saint-jean Languedoc, Toulouse